CLINICAL TRIAL: NCT00387465
Title: A Phase I/II Study of Entinostat in Combination With 5-Azacytidine in Patients With Recurrent Advanced Non-Small Cell Lung Cancer
Brief Title: Azacitidine and Entinostat in Treating Patients With Recurrent Advanced Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00220; NCI-2009-00220 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000504083 (Other: Clinical Data Repository); NA_00003114 (Other: Johns Hopkins IRB); J0658 (Other: SKCCC); 7759 (Other: CTEP); P30CA006973 (NIH); U01CA070095 (NIH)
Record Dates: First submitted 2006-10-12; First posted 2006-10-13 (Estimated); Results first posted 2019-05-09 (Actual); Last update posted 2019-05-09 (Actual); Status verified 2019-04

CONDITIONS: Recurrent Non-Small Cell Lung Carcinoma; Stage IIIA Non-Small Cell Lung Cancer; Stage IIIB Non-Small Cell Lung Cancer; Stage IV Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Azacitidine; entinostat

ARMS (3):
- Phase I - 30mg/m2 Azacitidine (Experimental): Patients receive Azacitidine 30mg/m2 SQ and entinostat 7mg PO on days 3 and 10 of each cycle.
  Interventions: Drug: Azacitidine 30mg/m2; Drug: Entinostat
- Phase I - 40mg/m2 Azacitidine (Experimental): Patients receive azacitidine 40mg/m2 SQ and entinostat 7mg PO on days 3 and 10 of each cycle.
  Interventions: Drug: Entinostat; Drug: Azacitidine 40mg/m2
- Phase II Arm (Experimental): Patients receive azacitidine 40mg/m2 subcutaneously (SQ) on days 1-6 and 8-10 and entinostat 7mg PO on days 3 and 10. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Entinostat; Drug: Azacitidine 40mg/m2

INTERVENTIONS:
Drug: Azacitidine 30mg/m2 — Azacitidine 30mg/m2 subcutaneously (SQ)
  Other Names: 5 AZC; 5-AC; 5-Azacytidine; 5-AZC; AZACITIDINE; Azacytidine; Azacytidine, 5-; Ladakamycin; Mylosar; U-18496; Vidaza
  Arms: Phase I - 30mg/m2 Azacitidine
Drug: Entinostat — 7mg by mouth (PO) on days 3 and 10 of each cycle
  Other Names: HDAC inhibitor SNDX-275; MS 27-275; MS-275; SNDX-275
Drug: Azacitidine 40mg/m2 — Azacitidine 40mg/m2 SQ
  Other Names: 5 AZC; 5-AC; 5-Azacytidine; 5-AZC; AZACITIDINE; Azacytidine; Azacytidine, 5-; Ladakamycin; Mylosar; U-18496; Vidaza
  Arms: Phase I - 40mg/m2 Azacitidine; Phase II Arm

SUMMARY:
This phase I/II trial is studying the side effects and best dose of azacitidine when given together with entinostat and to see how well they work in treating patients with recurrent advanced non-small cell lung cancer. Azacitidine and entinostat may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving azacitidine together with entinostat may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess safety, characterize toxicities, and determine the maximum tolerated dose of 5-AZA (azacitidine) with a fixed-dose of entinostat in patients with recurrent advanced non-small cell lung cancer (NSCLC). (Phase I) II. To determine the objective response rate of 5-AZA and entinostat in patients with recurrent NSCLC. (Phase II)

SECONDARY OBJECTIVES:

I. To determine the pharmacokinetic profile of 5-AZA and entinostat in patients with recurrent NSCLC.

II. To assess the pharmacodynamic effects of 5-AZA and entinostat on deoxyribonucleic acid (DNA) methylation, histone acetylation, and gene re-expression in patients with recurrent NSCLC through analysis of blood, sputum and tissue biopsies.

III. To explore the effect of 5-AZA and entinostat on progression-free and overall survival in patients with recurrent advanced non-small cell lung cancer.

IV. To explore the differing response rates and progression-free survivals of two schedules of 5-AZA and entinostat in patients with recurrent advanced non-small cell lung cancer.

OUTLINE: This is a multicenter, phase I, dose-escalation study of azacitidine followed by an open-label, phase II study.

Patients receive azacitidine subcutaneously (SC) on days 1-6 and 8-10 and entinostat orally (PO) on days 3 and 10. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed metastatic or unresectable NSCLC
* Patient must have failed at least one previous chemotherapy regimen
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as >= 20 mm with conventional techniques or as >= 10 mm with spiral computed tomography (CT) scan
* Life expectancy of greater than 12 weeks
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) =< 2 (Karnofsky >= 60%)
* Leukocytes >= 3,000/mcL
* Absolute neutrophil count >= 1,500/mcL
* Platelet count >= 100,000/mcL
* Total bilirubin within normal institutional limits
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT] and alanine aminotransferase (ALT) (serum glutamic pyruvate transaminase [SGPT]) =< 2.5 x upper limit of normal
* Creatinine within normal institutional limits OR creatinine clearance >= 60 mL/min/1.73m^2 for patients with creatinine levels above institutional normal
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Ability to understand and the willingness to sign a written informed consent document
* Patients who have a major objective response to treatment on this protocol, and who experience progression of disease at least 1 year after completion of protocol consent and therapy, may be re-treated at the previously effective dose and schedule

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier
* Patients may not be receiving any other investigational agents
* Patients with uncontrolled brain metastases; patients with brain metastases must have stable neurologic status following local therapy (surgery or radiation) for at least 4 weeks, and must be without neurologic dysfunction that would confound the evaluation of neurologic and other adverse events
* Patients with liver metastases that replace greater than 30% of the liver parenchyma
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to entinostat, 5-AZA, mannitol or other agents used in the study
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study; breastfeeding should be discontinued if the mother is treated on this protocol
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2006-08; Primary Completion 2014-05 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Wrangle, Principal Investigator — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins Hospital
Locations (5):
- United States (5):
  - USC Norris Comprehensive Cancer Center, Los Angeles, California
  - Sidney Kimmel Cancer Center, San Diego, California
  - Johns Hopkins Bayview Medical Center, Baltimore, Maryland
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins Hospital, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland

REFERENCES:
- [Result] Juergens RA, Wrangle J, Vendetti FP, Murphy SC, Zhao M, Coleman B, Sebree R, Rodgers K, Hooker CM, Franco N, Lee B, Tsai S, Delgado IE, Rudek MA, Belinsky SA, Herman JG, Baylin SB, Brock MV, Rudin CM. Combination epigenetic therapy has efficacy in patients with refractory advanced non-small cell lung cancer. Cancer Discov. 2011 Dec;1(7):598-607. doi: 10.1158/2159-8290.CD-11-0214. Epub 2011 Nov 9. PMID 22586682

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 49 subjects did not start the study due to screen failure or PI decision.
Period: Overall Study
Arm/Group | Phase I - 30mg/m2 Azacitidine | Phase I - 40mg/m2 Azacitidine | Phase II Arm
Started | 3 | 7 | 35
Completed | 3 | 6 | 35
Not Completed | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase II Arm | Phase I - 30mg/m2 Azacitidine | Phase I - 40mg/m2 Azacitidine | Total
Number analyzed (Participants) | 35 | 3 | 7 | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 18 | 3 | 4 | 25
  >=65 years | 17 | 0 | 3 | 20
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 0 | 4 | 22
  Male | 17 | 3 | 3 | 23
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 35 | 3 | 7 | 45

OUTCOME MEASURES:

1. Primary Outcome: (Phase I) Maximum Tolerated Dose (MTD) of Azacitidine When Given Together With Entinostat as Determined by Number of Participants Experiencing Dose-limiting Toxicity (DLT)
Description: DLT is defined by the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v3.0
Time Frame: Up to 28 days
Population: Only participants in the Phase I arms were analyzed for this outcome measure
Measure: Count of Participants; unit: Participants
Arm/Group | Phase II Arm | Phase I - 30mg/m2 Azacitidine | Phase I - 40mg/m2 Azacitidine
Number analyzed (Participants) | 0 | 3 | 6
Participants |  | 0 | 0
Statistical Analysis 1: Comparison: Phase I - 30mg/m2 Azacitidine vs Phase I - 40mg/m2 Azacitidine; Test type: Other — The maximum tolerated dose (MTD) was derived from the number of participants experiencing dose-limiting toxicities in the Phase I arms. The MTD was the dose at which ≤30% of patients experienced DLTs during cycle 1 up to a pre-specified maximal dose of 40 mg/m2 of azacitidine; Maximum Tolerated Dose = 40 — MTD of Azacitidine measured in mg/m^2

2. Primary Outcome: (Phase II) Objective Response Rate After Treatment With Azacitidine and Entinostat as Assessed by Number of Participants With Response After at Least One Cycle of Therapy
Description: Number of participants with progressive disease (PD), stable disease (SD), complete response (CR), or partial response (PR), as defined by Response Evaluation Criteria in Solid Tumors (RECIST 1.0), after completing at least one cycle of therapy. Per RECIST 1.0, progression is defined as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions; PR is defined as >=30% decrease in the sum of the longest diameter of target lesions, CR is defined as the disappearance of all target lesions.
Time Frame: Up to 8 years
Population: Only participants who received Azacitidine 40mg/m2 and completed at least one cycle of therapy were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Groups:
- Azacitidine 40mg/m2 With Entinostat: Patients receive azacitidine 40mg/m2 SC on days 1-6 and 8-10 and entinostat PO on days 3 and 10. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.
Arm/Group | Azacitidine 40mg/m2 With Entinostat
Number analyzed (Participants) | 34
Participants
  CR | 1
  PD | 22
  PR | 1
  SD | 10

3. Secondary Outcome: Effect of Entinostat and Azacitidine on DNA Methylation and Response
Description: Number of participants with decrease in DNA methylation ("methylation-signature positive") on Day 10 or Day 29, and either stable disease or objective response (OR) as defined by RECIST 1.0. Per RECIST 1.0, progression is defined as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions; PR is defined as >=30% decrease in the sum of the longest diameter of target lesions, complete response is defined as disappearance of all target lesions; OR=CR+PR.
Time Frame: Baseline and days 10 and 29
Population: Only participants who received Azacitidine 40mg/m2 (42 participants) were assessed for this outcome measure. Therefore, data was not collected from the participants in the 30mg/m2 arm from Phase I. However, data was evaluable in only 26/42 participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Azacitidine 40mg/m2 With Entinostat
Number analyzed (Participants) | 26
Participants | 8

4. Secondary Outcome: Major Objective Response After Immediate Subsequent Therapy as Measured by Number of Participants With PR, SD, PD After at Least 1 Cycle of Subsequent Chemotherapy
Description: Number of participants with progressive disease (PD), stable disease (SD), or partial response (PR), as defined by Response Evaluation Criteria in Solid Tumors (RECIST 1.0) after at least 1 cycle of subsequent chemotherapy. Per RECIST 1.0, progression is defined as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions; PR is defined as >=30% decrease in the sum of the longest diameter of target lesions.
Time Frame: Up to 8 years
Population: Only participants who received 40mg/m2 azacitidine and at least 1 cycle of subsequent chemotherapy (19 participants) were assessed for this outcome measure. Therefore, data was not collected from the participants in the 30mg/m2 arm from Phase I. However, 2/19 deceased prior to imaging and therefore were not evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Azacitidine 40mg/m2 With Entinostat
Number analyzed (Participants) | 17
Participants
  PR | 4
  SD | 9
  PD | 4

5. Secondary Outcome: Overall Survival
Description: Determined by the method determined by Kaplan and Meier. 95% confidence intervals will be estimated.
Time Frame: Up to 1 year
Population: Only participants who received Azacitidine 40mg/m2 were evaluable for this outcome measure.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Azacitidine 40mg/m2 With Entinostat
Number analyzed (Participants) | 42
months | 6.4 [3.8 to 9.2]

6. Secondary Outcome: Pharmacokinetic Profile of Azacytidine as Measured by Tmax
Description: Time to maximal concentration of azacitidine in the blood.
Time Frame: Day 1
Population: Only participants who received Azacitidine 40mg/m2 (42 participants) were assessed for this outcome measure. Therefore, data was not collected from the participants in the 30mg/m2 arm from Phase I. Data was not collected from 2/42 participants.
Measure: Median (Full Range); unit: hours
Arm/Group | Azacitidine 40mg/m2 With Entinostat
Number analyzed (Participants) | 40
hours | 0.5 [0.25 to 2.00]

7. Secondary Outcome: Progression-free Survival
Description: Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions. Determined by the method determined by Kaplan and Meier. 95% confidence intervals will be estimated.
Time Frame: Up to 1 year
Population: Only participants who received Azacitidine 40mg/m2 were assessed for this outcome measure. Therefore, data was not collected from the participants in the 30mg/m2 arm from Phase I.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Azacitidine 40mg/m2 With Entinostat
Number analyzed (Participants) | 42
weeks | 7.4 [7.0 to 8.0]

8. Secondary Outcome: Pharmacokinetic Profile of Azacitidine as Measured by Cmax
Description: Maximal concentration (ng/mL) of azacitidine
Time Frame: Day 1
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Azacitidine 40mg/m2 With Entinostat
Number analyzed (Participants) | 40
ng/mL | 468 (241)

9. Secondary Outcome: Pharmacokinetic Profile of Azacitidine as Measured by AUC (ng*hr/mL)
Time Frame: Day 1
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Azacitidine 40mg/m2 With Entinostat
Number analyzed (Participants) | 40
ng*hr/mL | 675 (290)

10. Secondary Outcome: Average Steady State Trough Concentration (ng/mL) of Entinostat
Time Frame: Day 10 and 17
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Azacitidine 40mg/m2 With Entinostat
Number analyzed (Participants) | 40
ng/mL
  Day 10 | 0.84 (0.23)
  Day 17 | 1.10 (0.34)

11. Secondary Outcome: Pharmacokinetic Profile of Azacitidine as Measured by Half-life
Time Frame: Day 1
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Azacitidine 40mg/m2 With Entinostat
Number analyzed (Participants) | 40
hours | 1.12 (1.06)

ADVERSE EVENTS:
Groups:
- Azacitidine 40mg/m2 and Entinostat: Patients from both Phase I and II who received azacitidine 40mg/m2 subcutaneously (SQ) on days 1-6 and 8-10 and entinostat 7mg PO on days 3 and 10. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.
Arm/Group | Azacitidine 40mg/m2 and Entinostat | Phase I - 30mg/m2 Azacitidine
All-Cause Mortality (participants affected / at risk) | 2/42 | 0/3
Serious Adverse Events (participants affected / at risk) | 2/42 | 0/3
Other Adverse Events (participants affected / at risk) | 36/42 | 0/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Azacitidine 40mg/m2 and Entinostat (N=42) | Phase I - 30mg/m2 Azacitidine (N=3)
Lymphopenia (Blood and lymphatic system disorders) | 2 | NA
Neutropenia (Blood and lymphatic system disorders) | 1 | NA
Pericardial Tamponade (Cardiac disorders) | 1 | NA
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Azacitidine 40mg/m2 and Entinostat (N=42) | Phase I - 30mg/m2 Azacitidine (N=3)
Anemia (Blood and lymphatic system disorders) | 20 | NA
Leukopenia (Blood and lymphatic system disorders) | 7 | NA
Lymphopenia (Blood and lymphatic system disorders) | 13 | NA
Neutropenai (Blood and lymphatic system disorders) | 3 | NA
Thrombocytopenia (Blood and lymphatic system disorders) | 5 | NA
Abdominal pain (Gastrointestinal disorders) | 6 | NA
Constipation (Gastrointestinal disorders) | 15 | NA
Diarrhea (Gastrointestinal disorders) | 7 | NA
Nausea (Gastrointestinal disorders) | 20 | NA
Vomiting (Gastrointestinal disorders) | 11 | NA
Hypokalemia (Metabolism and nutrition disorders) | 3 | NA
Hyponatremia (Metabolism and nutrition disorders) | 7 | NA
Anorexia (General disorders) | 16 | NA
Dyspnea (General disorders) | 9 | NA
Fatigue (General disorders) | 25 | NA
Chills (General disorders) | 1 | NA
Left chest pain (General disorders) | 1 | NA
Injection site reaction (General disorders) | 25 | NA
Urinary Tract infection (Renal and urinary disorders) | 1 | NA
Dizziness (General disorders) | 11 | NA
Hemmorhoids (General disorders) | 1 | NA
Blurred Vision (General disorders) | 2 | NA
Confusion (Psychiatric disorders) | 3 | NA
Preformance status decline (General disorders) | 1 | NA
Aphasia (General disorders) | 1 | NA
Pitting edema (Skin and subcutaneous tissue disorders) | 1 | NA
Hypotension (Cardiac disorders) | 7 | NA
Albumin (Hepatobiliary disorders) | 12 | NA
Alk Phos (Hepatobiliary disorders) | 9 | NA
AST (Hepatobiliary disorders) | 2 | NA
ALT (Hepatobiliary disorders) | 2 | NA
Bilirubin (Hepatobiliary disorders) | 3 | NA
Hyperglycemia (Metabolism and nutrition disorders) | 18 | NA
Hypomagnesemia (Metabolism and nutrition disorders) | 3 | NA
Cough (General disorders) | 2 | NA
Hypoxic (General disorders) | 1 | NA
Tachycardia (Cardiac disorders) | 3 | NA
Dehydration (Gastrointestinal disorders) | 3 | NA
Weight loss (Gastrointestinal disorders) | 5 | NA
Uric Acid (General disorders) | 1 | NA
Elevated creatinine (General disorders) | 5 | NA
Back pain (Musculoskeletal and connective tissue disorders) | 1 | NA
Inter. Muscle Spasm (Musculoskeletal and connective tissue disorders) | 1 | NA
Hyperkalemia (General disorders) | 1 | NA
Hypermagnesemia (General disorders) | 2 | NA
Heartburn (Cardiac disorders) | 2 | NA
Upset stomach (Gastrointestinal disorders) | 1 | NA
Insomnia (General disorders) | 4 | NA
Depression or Anxiety (Psychiatric disorders) | 5 | NA
Fever (General disorders) | 4 | NA
Hypercalcemia (Metabolism and nutrition disorders) | 1 | NA
Hypocalcemia (Metabolism and nutrition disorders) | 5 | NA
Somnolence (General disorders) | 1 | NA
Aches (General disorders) | 2 | NA
Hypophosphetemia (Metabolism and nutrition disorders) | 4 | NA
Throat Pain (General disorders) | 1 | NA
A.filbrillation (Cardiac disorders) | 1 | NA
GIB (General disorders) | 1 | NA
Weakness (General disorders) | 2 | NA
Pleural Effusion (General disorders) | 3 | NA
Headache (General disorders) | 3 | NA
Stroke (General disorders) | 1 | NA
Lung Infection (General disorders) | 2 | NA
Myositis (General disorders) | 1 | NA
Neuropathy (General disorders) | 1 | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less